CLINICAL TRIAL: NCT02061748
Title: The Comparative Safety and Effectiveness of Warfarin and Dabigatran Utilized in the Humana Non-Valvular Atrial Fibrillation (NVAF) Patient Population-A Retrospective Database Analysis
Brief Title: The Comparative Safety and Effectiveness of Warfarin and Dabigatran Prescribed in the Non-valvular Atrial Fibrillation Population With Humana Healthcare Coverage
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.192
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- dabigatran
  Interventions: Drug: Observational
- warfarin

INTERVENTIONS:
Drug: Observational — Retrospective Chart Review
  Groups: dabigatran

SUMMARY:
This study is an opportunity for Boehringer Ingelheim to collaborate with Humana to conduct comparative safety and effectiveness studies of dabigatran and warfarin using real world data from Humana's health plan operations.

DETAILED DESCRIPTION:
Study Design:

n/a

ELIGIBILITY:
Inclusion criteria:

* Patient must have at least one inpatient, one physician office visit, or one emergency room visit with a diagnosis of AF on the index date or during the pre-index period.
* Patients must be continuously enrolled in a health plan during the pre-index period
* Patient must have a prescription for dabigatran or warfarin
* Patient must be treatment naive from all oral anticoagulant (OAC) use prior to first OAC prescription
* Aged 18-89 years on the index date. The index date is defined as the date of the first OAC prescription

Exclusion criteria:

* Diagnosis of hyperthyroidism during the pre-index period,
* Having claims for any of the following within 3 months prior to the first diagnosis of AF: cardiac surgery, pericarditis, myocarditis, pulmonary embolism.
* Any patients with at least one medical claim for valvular heart disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF
Sampling Method: Non-Probability Sample
Enrollment: 38499 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Comprehensive Health Insights, Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-interventional study based on existing data was conducted. This is a retrospective database analysis to assess the safety and effectiveness of dabigatran compared to warfarin in patients diagnosed with non-valvular atrial fibrillation (NVAF) in the real-world setting using the Humana population.
Pre-assignment Details: Participant flow and demographic section is based on Pre-propensity score matching data however to analyze the outcome measures Post-propensity score matching data were used.
Groups:
- Dabigatran: Patients with ≥1 pharmacy claim for dabigatran between October 1, 2010 and April 30, 2013 were identified as dabigatran users. Patients received 75 or 150 milligram (mg) dabigatran capsules orally, twice daily.
- Warfarin: Patients with ≥1 pharmacy claim for warfarin between October 1, 2010 and April 30, 2013 were identified as warfarin users. Patients received 1 to 10 mg tablets, administered orally.
Period: Overall Study
Arm/Group | Dabigatran | Warfarin
Started | 7646 | 30853
Completed | 7646 | 30853
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of selected patients (total) before propensity score matching.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Total
Number analyzed (Participants) | 7646 | 30853 | 38499
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (8.6) | 74.8 (8.2) | 74.5 (8.3)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 3316 | 13944 | 17260
  Male | 4330 | 16906 | 21236
  Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stroke (Primary Analysis)
Description: This outcome measure describes the incidence of stroke (hemorrhagic and ischemic) for dabigatran and warfarin in the primary analysis.
  Ischemic stroke includes: Occlusion and stenosis of precerebral arteries with cerebral infarction, Occlusion of cerebral arteries with cerebral infarction and Acute, but ill-defined, cerebrovascular disease but excludes above diagnosis if hospitalization lasted less than 48 hours and was accompanied by carotid endarterectomy.
  Hemorrhagic stroke includes: Subarachnoid hemorrhage (SAH) and Intracerebral hemorrhage (ICH) but excludes previous listed diagnoses if "traumatic brain injury" or "rehabilitation care" is present.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: From 1 October 2010 to 30 April 2013 identified with index date (first prescription of dabigatran or warfarin) plus a follow-up period of 12 months (up to 42 months)
Population: A total of 7245 dabigatran and 14490 warfarin users remained after propensity score matching (PSM, 1:2) which was used to control for channelling bias.
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 21.9 [17.4 to 26.5] | 29.3 [25.7 to 32.9]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; Study outcomes for the primary analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization; Test type: Superiority or Other; p = 0.0111, Chi-squared

2. Primary Outcome: Stroke (Post-hoc Analysis)
Description: This outcome measure describes the incidence of stroke (hemorrhagic and ischemic) for dabigatran and warfarin in the post-hoc analysis. A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 12.4 [9.0 to 15.8] | 16.1 [13.4 to 18.7]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; The post-hoc analysis defined the principal diagnosis as the primary diagnosis on the first inpatient hospital claim with a room and board charge; Test type: Superiority or Other; p = 0.0861, Chi-squared

3. Primary Outcome: Major Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major bleeding (hemorrhagic stroke, major intracranial bleeding and major extracranial bleeding) for dabigatran and warfarin in the primary analysis.
  Major Intracranial Bleeding includes subarachnoid hemorrhage, intracerebral hemorrhage, other and unspecified intracranial hemorrhage, subarachnoid hemorrhage following injury without mention of open intracranial wound, subdural hemorrhage following injury without mention of open intracranial wound, extradural hemorrhage following injury without mention of open intracranial wound, other and unspecified intracranial hemorrhage following injury without mention of open intracranial wound but excludes these codes if major trauma was present. Major extracranial bleeding includes major gastrointestinal (GI) bleeding, major urogenital bleeding and major other bleeding. Either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization were used.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 61.7 [54.1 to 69.3] | 76.7 [70.9 to 82.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0011, Chi-squared

4. Primary Outcome: Major Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major bleeding (Inclusive of hemorrhagic stroke, major intracranial bleeding and major extracranial bleeding) for dabigatran and warfarin in the post-hoc analysis. A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 35.6 [29.8 to 41.4] | 46.9 [42.4 to 51.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0019, Chi-squared

5. Secondary Outcome: Ischemic Stroke (Primary Analysis)
Description: This outcome measure describes the incidence of ischemic stroke for dabigatran and warfarin in the primary analysis. Ischemic stroke includes: Occlusion and stenosis of precerebral arteries with cerebral infarction, Occlusion of cerebral arteries with cerebral infarction and Acute, but ill-defined, cerebrovascular disease but excludes above diagnosis if hospitalization lasted less than 48 hours and was accompanied by carotid endarterectomy.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 21.7 [17.2 to 26.2] | 26.4 [23.0 to 29.8]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0808, Chi-squared

6. Secondary Outcome: Ischemic Stroke (Post-hoc Analysis)
Description: This outcome measure describes the incidence of ischemic stroke for dabigatran and warfarin in the post-hoc analysis. Ischemic stroke includes: Occlusion and stenosis of precerebral arteries with cerebral infarction, Occlusion of cerebral arteries with cerebral infarction and Acute, but ill-defined, cerebrovascular disease but excludes above diagnosis if hospitalization lasted less than 48 hours and was accompanied by carotid endarterectomy.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 11.2 [8.0 to 14.5] | 12.9 [10.6 to 15.3]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3502, Chi-squared

7. Secondary Outcome: Hemorrhagic Stroke (Primary Analysis)
Description: This outcome measure describes the incidence of hemorrhagic stroke for dabigatran and warfarin in the primary analysis. Hemorrhagic stroke includes: subarachnoid hemorrhage, intracerebral hemorrhage but excludes these codes if "traumatic brain injury" or "rehabilitation care" as primary code is present.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 1.5 [0.3 to 2.6] | 4.4 [3.0 to 5.8]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0068, Chi-squared

8. Secondary Outcome: Hemorrhagic Stroke (Post-hoc Analysis)
Description: This outcome measure describes the incidence of hemorrhagic stroke for dabigatran and warfarin in the post-hoc analysis. Hemorrhagic stroke includes: Subarachnoid hemorrhage and intracerebral hemorrhage but excludes these codes if "traumatic brain injury" or "rehabilitation care" as primary code is present.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 1.2 [0.2 to 2.3] | 3.3 [2.1 to 4.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0271, Chi-squared

9. Secondary Outcome: Major Intracranial Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major intracranial bleeding for dabigatran and warfarin in the primary analysis. Major intracranial bleeding includes: Subarachnoid hemorrhage, intracerebral hemorrhage, other and unspecified intracranial hemorrhage, subarachnoid, subdural or extradural hemorrhage following injury without mention of open intracranial wound other and unspecified intracranial hemorrhage following injury without mention of open intracranial wound but excludes these codes if concomitant discharge diagnosis of major trauma was present.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 8.0 [5.3 to 10.8] | 11.3 [9.1 to 13.6]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0749, Chi-squared

10. Secondary Outcome: Major Intracranial Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major intracranial bleeding for dabigatran and warfarin in the post-hoc analysis. Major intracranial bleeding includes: Subarachnoid hemorrhage, intracerebral hemorrhage, other and unspecified intracranial hemorrhage, subarachnoid, subdural or extradural hemorrhage following injury without mention of open intracranial wound other and unspecified intracranial hemorrhage following injury without mention of open intracranial wound but excludes these codes if concomitant discharge diagnosis of major trauma was present.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 4.4 [2.4 to 6.4] | 8.6 [6.7 to 10.6]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0072, Chi-squared

11. Secondary Outcome: Major Extracranial Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major extracranial bleeding for dabigatran and warfarin in the primary analysis. Major extracranial bleeding includes: major gastrointestinal (GI) bleeding, major urogenital bleeding and major other bleeding.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 54.4 [47.2 to 61.5] | 66.1 [60.8 to 71.5]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0055, Chi-squared

12. Secondary Outcome: Major Extracranial Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major extracranial bleeding for dabigatran and warfarin in the post-hoc analysis. Major extracranial bleeding includes: major gastrointestinal (GI) bleeding, major urogenital bleeding and major other bleeding.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 31.2 [25.8 to 36.6] | 38.3 [34.2 to 42.3]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0284, Chi-squared

13. Secondary Outcome: Major GI Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major GI bleeding for dabigatran and warfarin in the primary analysis. Major GI bleeding includes major upper GI bleeding and major lower GI bleeding.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 44.4 [37.9 to 50.8] | 44.0 [39.7 to 48.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.907, Chi-squared

14. Secondary Outcome: Major GI Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major GI bleeding for dabigatran and warfarin in the post-hoc analysis. Major GI bleeding includes major upper GI bleeding and major lower GI bleeding.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 28.5 [23.4 to 33.7] | 28.7 [25.2 to 32.2]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8208, Chi-squared

15. Secondary Outcome: Major Upper GI Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major upper GI bleeding for dabigatran and warfarin in the primary analysis. Major upper GI bleeding includes acute gastric ulcer, chronic or unspecified gastric ulcer, acute duodenal ulcer, chronic or unspecified duodenal ulcer, acute, chronic or unspecified peptic ulcer, acute gastrojejunal ulcer, chronic or unspecified gastrojejunal ulcer with hemorrhage with/without obstruction and with hemorrhage and perforation with/without obstruction, hematemesis, endoscopic control of gastric or duodenal bleeding, upper gastrointestinal endoscopy including esophagus, stomach, and either the duodenum and/or jejunum as appropriate with control of bleeding, any method. Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 6.6 [4.1 to 9.1] | 9.0 [7.0 to 10.9]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1534, Chi-squared

16. Secondary Outcome: Major Upper GI Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major upper GI bleeding for dabigatran and warfarin in the post-hoc analysis. Major upper GI bleeding includes acute, chronic or unspecified gastric ulcer, acute duodenal ulcer, chronic or unspecified duodenal ulcer, acute, chronic or unspecified peptic ulcer, acute, chronic or unspecified gastrojejunal ulcer with hemorrhage with/without (w/wo) obstruction and with hemorrhage and perforation w/wo obstruction, hematemesis, endoscopic control of gastric or duodenal bleeding, upper gastrointestinal endoscopy including esophagus, stomach, and either the duodenum and/or jejunum as appropriate with control of bleeding, any method. A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. This was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 5.4 [3.1 to 7.6] | 6.8 [5.1 to 8.6]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3055, Chi-squared

17. Secondary Outcome: Major Lower GI Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major lower GI bleeding for dabigatran and warfarin in the primary analysis. Major lower GI bleeding includes diverticulosis or diverticulitis of small intestine or of colon with hemorrhage, hemorrhage of rectum and anus, angiodysplasia of intestine with hemorrhage, blood in stool and hemorrhage of GI tract (unspecified).
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 43.4 [37.0 to 49.8] | 42.8 [38.5 to 47.1]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9573, Chi-squared

18. Secondary Outcome: Major Lower GI Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major lower GI bleeding for dabigatran and warfarin in the post-hoc analysis.
  Major lower GI bleeding includes diverticulosis or diverticulitis of small intestine or of colon with hemorrhage, hemorrhage of rectum and anus, angiodysplasia of intestine with hemorrhage, blood in stool and hemorrhage of GI tract (unspecified).
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 23.6 [18.9 to 28.3] | 22.7 [19.6 to 25.8]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8465, Chi-squared

19. Secondary Outcome: Major Urogenital Bleeding (Primary Analysis)
Description: This outcome measure describes the incidence of major urogenital bleeding for dabigatran and warfarin in the primary analysis. Major urogenital bleeding includes hematuria and excessive/frequent menstruation and secondary diagnosis indicating acute bleeding (anemia).
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 5.8 [3.5 to 8.2] | 12.1 [9.8 to 14.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, Chi-squared

20. Secondary Outcome: Major Urogenital Bleeding (Post-hoc Analysis)
Description: This outcome measure describes the incidence of major urogenital bleeding for dabigatran and warfarin in the post-hoc analysis.
  Major urogenital bleeding includes hematuria and excessive/frequent menstruation and secondary diagnosis indicating acute bleeding (anemia).
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 0.2 [0.0 to 0.7] | 4.5 [3.1 to 5.9]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared

21. Secondary Outcome: Other Major Bleeds (Primary Analysis)
Description: This outcome measure describes the incidence of other major bleeds for dabigatran and warfarin in the primary analysis. Other major bleeds includes hemarthrosis, hemopericardium, hemoptysis, epistaxis, hemorrhage (not specified) and acute posthemorrhagic anemia.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 12.7 [9.2 to 16.1] | 18.2 [15.4 to 21.0]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0185, Chi-squared

22. Secondary Outcome: Other Major Bleeds (Post-hoc Analysis)
Description: This outcome measure describes the incidence of other major bleeds for dabigatran and warfarin in the post-hoc analysis.
  Other major bleeds includes hemarthrosis, hemopericardium, hemoptysis, epistaxis, hemorrhage (not specified) and acute posthemorrhagic anemia.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 2.7 [1.1 to 4.3] | 5.8 [4.3 to 7.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0138, Chi-squared

23. Secondary Outcome: Transient Ischemic Attack (TIA) (Primary Analysis)
Description: This outcome measure describes the incidence of TIA for dabigatran and warfarin in the primary analysis. TIA includes transient cerebral ischemia as the principal (primary) discharge diagnosis.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 10.7 [7.6 to 13.9] | 13.0 [10.7 to 15.4]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.261, Chi-squared

24. Secondary Outcome: TIA (Post-hoc Analysis)
Description: This outcome measure describes the incidence of TIA for dabigatran and warfarin in the post-hoc analysis.
  TIA includes transient cerebral ischemia as the principal (primary) discharge diagnosis.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 3.4 [1.6 to 5.2] | 4.4 [3.0 to 5.8]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4407, Chi-squared

25. Secondary Outcome: Myocardial Infarction (MI) (Primary Analysis)
Description: This outcome measure describes the incidence of MI for dabigatran and warfarin in the primary analysis. MI includes the acute myocardial infarction. Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 13.6 [10.1 to 17.2] | 16.1 [13.4 to 18.7]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2665, Chi-squared

26. Secondary Outcome: MI (Post-hoc Analysis)
Description: This outcome measure describes the incidence of MI for dabigatran and warfarin in the post-hoc analysis.
  MI includes the acute myocardial infarction. A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 8.0 [5.3 to 10.8] | 7.5 [5.7 to 9.3]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8017, Chi-squared

27. Secondary Outcome: Venous Thromboembolism (Primary Analysis)
Description: This outcome measure describes the incidence of venous thromboembolism for dabigatran and warfarin in the primary analysis. Venous thromboembolism includes the deep vein thrombosis and the pulmonary embolism.
  Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 12.2 [8.8 to 15.6] | 23.0 [19.9 to 26.2]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared

28. Secondary Outcome: Venous Thromboembolism (Post-hoc Analysis)
Description: This outcome measure describes the incidence of venous thromboembolism for dabigatran and warfarin in the post-hoc analysis.
  Venous thromboembolism includes the deep vein thrombosis and the pulmonary embolism.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 2.2 [0.8 to 3.6] | 3.5 [2.3 to 4.7]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2083, Chi-squared

29. Secondary Outcome: Deep Vein Thrombosis (Primary Analysis)
Description: This outcome measure describes the incidence of deep vein thrombosis for dabigatran and warfarin in the primary analysis. Deep vein thrombosis includes phlebitis and thrombophlebitis and other venous embolism and thrombosis. Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 9.5 [6.5 to 12.5] | 15.9 [13.3 to 18.6]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0023, Chi-squared

30. Secondary Outcome: Deep Vein Thrombosis (Post-hoc Analysis)
Description: This outcome measure describes the incidence of deep vein thrombosis for dabigatran and warfarin in the post-hoc analysis.
  Deep vein thrombosis includes phlebitis and thrombophlebitis and other venous embolism and thrombosis.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 1.0 [0.0 to 1.9] | 1.3 [0.6 to 2.1]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5331, Chi-squared

31. Secondary Outcome: Pulmonary Embolism (Primary Analysis)
Description: This outcome measure describes the incidence of pulmonary embolism for dabigatran and warfarin in the primary analysis. Pulmonary embolism includes acute pulmonary heart disease. Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 3.4 [1.6 to 5.2] | 9.1 [7.1 to 11.1]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, Chi-squared

32. Secondary Outcome: Pulmonary Embolism (Post-hoc Analysis)
Description: This outcome measure describes the incidence of pulmonary embolism for dabigatran and warfarin in the post-hoc analysis.
  Pulmonary embolism includes acute pulmonary heart disease. A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 1.2 [0.2 to 2.3] | 2.1 [1.2 to 3.1]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2646, Chi-squared

33. Secondary Outcome: All-cause Death (Primary Analysis)
Description: This outcome measure describes the incidence of death for dabigatran and warfarin in the primary analysis. Study outcomes for this analysis were identified using either the admitting diagnoses or on any of the service lines associated with an inpatient hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 36.6 [30.7 to 42.4] | 49.8 [45.2 to 54.5]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, Chi-squared

34. Secondary Outcome: All-cause Death (Post-hoc Analysis)
Description: This outcome measure describes the incidence of death for dabigatran and warfarin in the post-hoc analysis.
  A post-hoc analysis was conducted that measured outcomes using an algorithm to define the principal diagnosis. The principal diagnosis was defined as the primary diagnosis on the first room and board charge record within a hospital admission. This method results in identification of a single outcome for a hospitalization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 patient-years
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 7245 | 14490
Events per 1000 patient-years | 36.6 [30.7 to 42.4] | 49.8 [45.2 to 54.5]
Statistical Analysis 1: Comparison: Dabigatran vs Warfarin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0004, Chi-squared

ADVERSE EVENTS:
Description: This is a retrospective, non-interventional study. Adverse events (other than the primary and secondary endpoints) were not collected per protocol. Number of patients in this adverse event tables set to "0" as not applicable is technically not possible.
Arm/Group | Dabigatran | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was retrospective study using the Humana database. Adverse events (other than the primary and secondary endpoints) were not collected per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.